CLINICAL TRIAL: NCT04978298
Title: A Phase 1, Randomized, Double-blind, Placebo- and Positive-controlled Study to Evaluate the Effect of Ozanimod on Pressor Response to Oral Tyramine in Healthy Adult Subjects
Brief Title: Study to Evaluate the Pressor Effect of Oral Tyramine During Ozanimod Treatment in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RPC-1063-CP-005
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Phase 1
MeSH Terms: interventions — Phenelzine; ozanimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Rasagiline group (Experimental): Participants will receive rasagiline once daily (QD) for 14 days from Days 59 to 72.
  Interventions: Other: Placebo; Drug: Rasigiline
- Phenelzine group (Experimental): Participants will receive phenelzine twice daily (BID) for 14 days from Days 59 to 72.
  Interventions: Other: Placebo; Drug: Phenelzine
- Ozanimod Therapeutic group (Experimental): Participants will receive ozanimod QD for 65 days (including the initial 7-day dose escalation) from Days 8 to 72.
  Interventions: Other: Placebo; Drug: Ozanimod
- Ozanimod Supra-therapeutic group (Experimental): Participants will receive ozanimod QD for 65 days (including the initial 10-day dose escalation) from Days 8 to 72.
  Interventions: Other: Placebo; Drug: Ozanimod
- Placebo (Placebo Comparator): Participants will receive matched appropriate placebos from Days 8 to 72.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo
Drug: Rasigiline — Rasigiline
  Arms: Rasagiline group
Drug: Phenelzine — Phenelzine
  Arms: Phenelzine group
Drug: Ozanimod — Ozanimod
  Arms: Ozanimod Supra-therapeutic group; Ozanimod Therapeutic group

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, active-controlled, comparator controlled, multi-dose, parallel-group study divided into three treatment periods and a follow-up period with five treatment groups. This study will be conducted at 1 clinical research unit (CRU) in the United States (US).

Period 1 will consist of daily escalating doses of tyramine administered until tyramine pressor response (defined as the tyramine dose required to increase systolic blood pressure by at least 30 mm Hg from the daily defined baseline in 3 consecutive measurements within 4 hours after tyramine dosing) is achieved or Day 7.

Participants who achieve tyramine pressor response at tyramine doses >/= 200mg and </= 700mg are eligible for continuation into Period 2 and will be randomized accordingly.

Depending on the group to which a participant is randomized, participants will receive rasagiline, phenelzine, ozanimod (therapeutic dose), ozanimod (supra-therapeutic dose), or placebo in Period 2. The duration of dosing depends on the group to which a participant is randomized.

In Period 3, all participants will undergo a sham tyramine challenge and receive a single dose of tyramine placebo. Participants who do not achieve tyramine pressor response following the sham challenge will continue with the tyramine challenge (ie, tyramine pressor tests) for up to 12 additional days.

Participants who receive at least one dose of study drug in Period 2 will participate in a follow-up phase during which 2 follow-up telephone calls will be performed, the last of which will occur approximately 80 to 100 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. Be a male or non-pregnant, non-lactating female, 25 to 55 years of age, inclusive, at the time of signing the informed consent form.
2. Must understand and voluntarily sign an informed consent form prior to any study-related assessments/procedures being conducted.
3. Is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Female participant must meet at least 1 of the following criteria:

   * Have a negative serum pregnancy test at Screening and Day -1 (females of child-bearing potential only).
   * Be postmenopausal (defined as 2 years after the last period and follicle-stimulating hormone > 40 IU/L).
   * Have received surgical sterilization (eg, bilateral tubal ligation, bilateral oophorectomy, hysterectomy) at least 6 months before Screening.
5. Female of child-bearing potential:

   Must agree to practice a highly effective method of contraception at least 28 days prior to first dose of investigational product until completion of the 90-day safety follow-up period. Highly effective methods of contraception are those that alone or in combination result in a failure rate of a Pearl index of less than 1% per year when used consistently and correctly.

   Examples of acceptable methods of birth control in this study are the following:
   * Combined hormonal (estrogen and progestogen containing) contraception, which may be oral, intravaginal, or transdermal
   * Progestogen-only hormonal contraception associated with inhibition of ovulation, which may be oral, injectable, or implantable
   * Placement of an intrauterine device or intrauterine hormone-releasing system
   * Bilateral tubal occlusion
   * Vasectomised partner
   * Complete sexual abstinence Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhoea method are not acceptable methods of contraception. Female condom and male condom should not be used together.
6. Has a body weight of at least 110 pounds (50 kg); body mass index within the range of 18.0 to 30.0 kg/m2, inclusive.
7. Is in good health, as determined by no clinically significant findings from medical or surgical history, 12-lead ECG, PE, clinical laboratory safety tests, and vital signs.
8. Has a mean systolic blood pressure (SBP) of 90 to 139 mm Hg, a diastolic blood pressure (DBP) of 50 to 89 mm Hg from three consecutive measurements at Screening and Day -1.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. an unstable SBP (ie, SBP exceeds a maximum range of 15 mm Hg between the lowest and highest values in three consecutive measurements within 15 minutes during Screening).
2. the presence or history of any clinically relevant abnormality, condition, or disease (such as glaucoma, liver disease or abnormal liver function tests, cardiovascular or pulmonary diseases) that, in the opinion of the Investigator, may affect absorption, distribution, metabolism, or elimination of the IPs, that would prevent the participant from participating in the study, or which places the participant at unacceptable risk if he/she were to participate in the study.
3. any condition that confounds the ability to interpret data from the study.
4. history of bipolar, depression or suicidal ideation or behavior, or a history of psychiatric illnesses.
5. history of clinically significant or unstable vascular disease, a history of syncope associated with hypotension within the last 2 years, a history of orthostatic hypotension (ie, SBP decrease of > 20 mm Hg between 2 and 5 minutes after standing compared with supine SBP), or a history of tachycardia or hypertension.
6. an estimated glomerular filtration rate (eGFR) < 80 mL/min/1.73 m2 according to the 2009 chronic kidney disease (CKD) epidemiology collaboration (CKD EPI) equation: eGFR = 141 × min(Scr/κ, 1) × max(Scr/κ, 1)-1.209 × 0.993Age × 1.018 [if female] × 1.159 [if African American] where: Scr is serum creatinine in mg/dL, κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/κ or 1, and max indicates the maximum of Scr/κ or 1.
7. a seated heart rate outside 55 to 95 beats per minute at Screening or Day -1.
8. a resting QTcF > 450 msec (males) or > 470 msec (females) or PR interval > 210 msec at Screening or Day -1 or at additional risk for QT interval prolongation.
9. a history of diabetes mellitus type 1, or uncontrolled diabetes mellitus type 2 with hemoglobin A1c (HbA1c) > 8%.
10. a history of uveitis (within the last year prior to Screening) or clinically confirmed diagnosis of macular edema.
11. a history of alcoholism, drug abuse, or addiction within 24 months prior to Screening.
12. a known active bacterial, viral, fungal (excluding fungal infection of nail beds, minor upper respiratory tract infections, and minor skin infections), mycobacterial infection (including tuberculosis or atypical mycobacterial disease) or any major episode of infection that required hospitalization or treatment with intravenous antibiotics within 30 days of Screening or oral antibiotics within 14 days of Screening.

    * In the case of prior SARS-CoV-2 infection, symptoms must have completely resolved and based on Investigator assessment in consultation with the Medical Monitor, there are no sequelae that would place the participant at a higher risk of receiving investigational treatment.
13. a positive serum test for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus .
14. used any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, electronic cigarettes, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 3 months prior to the first dose of IP.
15. consumed marijuana products within 3 months prior to the first dose of IP.
16. a positive urine drug test including cotinine at Screening or Day -1.
17. a positive alcohol breath or urine test at Screening or Day -1.
18. received any investigational drug within 30 days or 5 times the elimination half-life (if known), whichever is longer, prior to the first dose of IP.
19. received a live or live attenuated vaccine within 4 weeks prior to the first dose of IP.
20. used any over-the-counter medication (excluding acetaminophen up to 1 g/day), dietary or herbal supplement (excluding vitamins/multi-vitamins), octopamine within 14 days prior to the first dose of IP. St. John's wort must be discontinued at least 28 days prior to the first dose of IP.
21. used any systemic prescription medication (excluding hormonal contraceptives) within 28 days or 5 times the elimination half-life, whichever is longer, prior to the first dose of IP.
22. used any MAO inhibitors within 90 days prior to the first dose of IP.
23. a history of allergic reaction to tyramine, phenelzine, rasagiline, or S1P agonist.
24. a history of adverse reactions to tyramine-containing foods.
25. ingested alcohol within 7 days prior to the first dose of IP.
26. fails or is unwilling to abstain from strenuous physical activities for at least 24 hours prior to the first dose of IP.
27. poor peripheral venous access.
28. donated greater than 400 mL of blood within 60 days prior to Day 1.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-02-26 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Tyramine Sensitivity Factor (TSF) | Up to Day 85
  The ratio of Tyramine pressor response (Tyr30) in Period 1 over Tyr30 in Period 3.

SECONDARY OUTCOMES:
Heart Rate (HR) | Up to Day 85
  Will be summarized descriptively by period, treatment group, day, and nominal time (where appropriate) using the per protocol (PP) population.
Systolic Blood Pressure (SBP) | Up to Day 85
  Will be summarized descriptively by period, treatment group, day, and nominal time (where appropriate) using the per protocol (PP) population.
Diastolic Blood Pressure (DBP) | Up to Day 85
  Will be summarized descriptively by period, treatment group, day, and nominal time (where appropriate) using the per protocol (PP) population.
CC112273 Pharmacokinetics: Cmax | Up to Day 85
  Maximum observed plasma concentration within the dosing interval.
CC112273 Pharmacokinetics: Cmin | Up to Day 85
  Minimum observed plasma concentration within the dosing interval.
CC112273 Pharmacokinetics: Tmax | Up to Day 85
  Time to Cmax.
CC112273 Pharmacokinetics: AUC0-24 | Up to Day 85
  Area under the concentration-time curve from time 0 to 24 hours.
CC112273 Pharmacokinetics: Ctrough | Up to Day 85
  Predose or trough concentration.
CC1084037 Pharmacokinetics: Cmax | Up to Day 85
  Maximum observed plasma concentration within the dosing interval.
CC1084037 Pharmacokinetics: Cmin | Up to Day 85
  Minimum observed plasma concentration within the dosing interval.
CC1084037 Pharmacokinetics: Tmax | Up to Day 85
  Time to Cmax.
CC1084037 Pharmacokinetics: AUC0-24 | Up to Day 85
  Area under the concentration-time curve from time 0 to 24 hours.
CC1084037 Pharmacokinetics: Ctrough | Up to Day 85
  Predose or trough concentration.
Ozanimod Pharmacokinetics: Cmax | Up to Day 85
  Maximum observed plasma concentration within the dosing interval.
Ozanimod Pharmacokinetics: Cmin | Up to Day 85
  Minimum observed plasma concentration within the dosing interval.
Ozanimod Pharmacokinetics: Tmax | Up to Day 85
  Time to Cmax.
Ozanimod Pharmacokinetics: AUC0-24 | Up to Day 85
  Area under the concentration-time curve from time 0 to 24 hours.
Ozanimod Pharmacokinetics: Ctrough | Up to Day 85
  Predose or trough concentration.
Pharmacokinetics for tyramine: Cave | Up to Day 85
  Average observed plasma concentration within the dosing interval.
Incidence of Adverse Events (AEs) | From screening until at least 90 days after last dose of study treatment (except for participants who discontinue from the study during Period 1 in which case AEs will be recorded from screening until 24 hours after the last dose of tyramine)
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a participant during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the participant's health, including laboratory test values regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Attanasio, MD, Study Director — Celgene
Locations (1):
- Local Institution - 001, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm